CLINICAL TRIAL: NCT05389527
Title: Efficacy and Safety of the Combination of Pembrolizumab and Lenvatinib as Neoadjuvant Treatment for Hepatocellular Carcinoma Patients
Brief Title: Pembrolizumab and Lenvatinib for Resectable Hepatocellular Carcinoma
Acronym: NeoLeap-HCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Hui-Chuan Sun, Professor of Surgery, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoLeap-HCC
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Neoadjuvant therapy; Pembrolizumab; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): Pembrolizumab+Lenvatinib
  Interventions: Drug: Pembrolizumab+Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab+Lenvatinib — After enrollment, subjects receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for 9 weeks: Lenvatinib 8 mg (body weight <60 kg) or 12 mg (body weight ≥60 kg) orally once daily for 9 weeks.
  Subjects conduct surgery 1 week after the last dose of Lenvatinib. 4 weeks after surgery, Pembrolizumab and Lenvatinib will restart as adjuvant treatment for up to 1 year.

SUMMARY:
This is an open-label, multi-center, single-arm, phase II study to evaluate the efficacy and safety of lenvatinib in combination with pembrolizumab as a neoadjuvant therapy in subjects with resectable hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The recurrence rate of hepatocellular carcinoma (HCC) after curative surgery is high and the survival benefit is limited. Neoadjuvant therapy, by targeting the disseminated tumor cells before curative surgery, may lower the incidence of tumor recurrence. In KEYNOTE-524 study, lenvatinib plus pembrolizumab combination showed promising efficacy and manageable toxicity. This study will evaluate the efficacy and safety of lenvatinib in combination with pembrolizumab as a neoadjuvant therapy in subjects with resectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically/cytologically or clinically (according to American Association for the Study of Liver Diseases (AASLD) criteria) confirmed diagnosis of HCC, excluding fibrolamellar sarcomatoid or mixed cholangiocarcinoma-hepatocellular carcinoma.
2. Have not received any locoregional or systemic treatment before enrolment. Patients had recurrence for more than 2 years after the previous surgery could be included.
3. Tumor within Milan criteria should be accompanied with microvascular invasion (judged by radionics nomogram of Fudan Zhongshan Hosp); Or beyond Milan criteria without extrahepatic metastasis.
4. Resectable disease as judged by a multidisciplinary treatment group.
5. Child-Pugh A.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 1 and performed within 7 days prior to date of enrolment.
7. In case of hepatitis B virus (HBV) positive (HBsAg (+)) subjects:

   * HBV DNA < 2000 IU/mL within 28 days before treatment; subjects received anti-HBV therapy should stay on the same therapy throughout study treatment.
   * Subjects with HBV DNA > 2000 IU/mL without anti-HBV therapy, should receive anti-HBV therapy and stay the same therapy throughout study treatment, and 2 days before treatment, the HBV DNA should decrease for at least 1 log.
   * Subjects with HBV DNA > 2000 IU/mL with anti-HBV therapy, should receive anti-HBV therapy and stay the same therapy throughout study treatment, and 2 days before treatment, the HBV DNA should decrease at least 1 log.
8. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mmHg at Screening and no change in antihypertensive medications within 1 week prior to the treatment.
9. Have measurable disease based on RECIST 1.1.
10. Have adequate organ function. Specimens collected within 7 days prior to start of study treatment.
11. Male participants: A male participant must agree to use a contraception of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
12. Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
13. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

Exclusion Criteria:

1. Imaging findings for HCC of clear invasion into the bile duct or portal vein invasion with Vp4.
2. Positive pregnancy test in female patients with childbearing potential within 72 hours prior to enrollment.
3. Prior anticancer treatment or any investigational agent.
4. Subjects having ≥2+ proteinuria on urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria. Subjects with urine protein ≥1 g/24-hour will be ineligible.
5. Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
6. New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months.
7. Prolongation of corrected QT (QTc , Fridericia formula) interval to >480 ms.
8. Gastrointestinal bleeding event or active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
9. Bleeding or thrombotic disorders or use of factor X inhibitors or anticoagulants requiring therapeutic international normalized ratio (INR) monitoring, eg, warfarin or similar agents. Treatment with low molecular weight heparin is permitted. Antiplatelet agents are prohibited throughout the study.
10. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
11. Subject is known to be positive for Human Immunodeficiency Virus (HIV).
12. Serious nonhealing wound, ulcer, or bone fracture.
13. History of solid organ or hematologic transplant.
14. Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial.
15. Active, known or suspected autoimmune disease that has required systemic treatment in the past 2 years or a documented history of clinically severe autoimmune disease, or any other syndrome that requires systemic steroids or immunosuppressive agents, patients with hypothyroidism stable on hormone replacement, or type 1 diabetes on insulin replacement will not be excluded from the study.
16. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis or has a history of interstitial lung disease.
17. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) | up to 24 weeks
  Defined as ≤ 50% viable tumor cells pathologically in the resected specimen.

SECONDARY OUTCOMES:
Pathologic complete response (pCR) | up to 24 weeks
  Defined as complete absence of residual visible tumor in resected tissues.
Objective response rate (ORR) | up to 24 weeks
  Defined as the proportion of the subjects who have a complete response (CR) and partial response (PR) per RECIST 1.1 in enrolled subjects
R0 resection rate | up to 24 weeks
  Defined as the proportion of patients who have microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed in enrolled subjects.
Disease-free survival (DFS) | up to 2 years
  Defined as the time from surgery to first documented recurrence or death due to any cause, whichever occurs first based on RECIST 1.1 in population underwent surgery
1-year DFS rate | up to 2 years
  Defined as the estimated proportion of patients who have no recurrence or death at 1 year after liver resection.
Overall survival | up to 2 years
  Defined as the time from enrollment to death due to any cause in enrolled subjects.
Adverse event (AE) | up to 2 years
  Adverse events (AEs) ; serious adverse events (SAEs); abnormal value of Lab test according to NCI-CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Huichuan Sun, Principal Investigator — Fudan University
Locations (4):
- China (4):
  - Zhongshan hospital, Shanghai, Shanghai Municipality
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - The first affiliated hospital, Yat-sen university, Guangzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Result] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739
- [Result] Pinato DJ, Fessas P, Sapisochin G, Marron TU. Perspectives on the Neoadjuvant Use of Immunotherapy in Hepatocellular Carcinoma. Hepatology. 2021 Jul;74(1):483-490. doi: 10.1002/hep.31697. Epub 2021 Jun 28. No abstract available. PMID 33369758